CLINICAL TRIAL: NCT01180322
Title: Randomized Phase-II Trial Evaluating Induction Therapy With Idarubicin and Etoposide Plus Sequential or Concurrent Azacitidine and Maintenance Therapy With Azacitidine
Brief Title: Trial Evaluating Induction Therapy With Idarubicin and Etoposide Plus Sequential or Concurrent Azacitidine and Maintenance Therapy With Azacitidine
Acronym: azacitidine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard Schlenk, PD Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 12-09
Record Dates: First submitted 2010-08-02; First posted 2010-08-12 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: azacitidine; Acute myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Etoposide; Azacitidine; Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Active Comparator): Standard Therapy
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: Lenograstim
- Arm B (Experimental): Investigational Therapy "Azacitidine Prior"
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: Azacitidine; Drug: Lenograstim
- Arm C (Experimental): Investigational Therapy "Azacitidine Concurrent"
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: Azacitidine; Drug: Lenograstim
- Arm D (Experimental): Investigational Therapy "Azacitidine After"
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Etoposide; Drug: Azacitidine; Drug: Lenograstim

INTERVENTIONS:
Drug: Cytarabine — Induction therapy:100 mg/m2/day by continuous intravenous (IV) infusion on days 1-7 (total dose 700 mg/m2)
  Consolidation therapy:
  Younger adults (18 to 65 years): 3 g/m2/day by IV infusion over 3 hours every 12 hours on days 1, 2, and 3 (total dose 18 g/m2).
  Elderly patients (>65 years): 1 g/m2/day by IV infusion over 3 hours every 12 hours on days 1, 2, and 3 (total dose 6 g/m2).
Drug: Idarubicin — First induction therapy:
  Arm A, C, D:
  12 mg/m2/day by IV push on days 1,3,5 (total dose 36 mg/m2). For elderly (>65 yrs) patients only two doses of idarubicin are foreseen on days 1+3.
  Arm B:
  12 mg/m2/day by IV push on days 6, 8 10 (total dose 36 mg/m2). For elderly (>65 yrs) patients only two doses of idarubicin are foreseen on days 6+8.
  Second induction therapy:
  Arm A, C, D:
  12 mg/m2/day by IV push on days 1 and 3 (total dose 24 mg/m2; for all age groups)
  Arm B:
  12 mg/m2/day by IV push on days 6 and 8 (total dose 24 mg/m2; for all age groups).
Drug: Etoposide — Induction therapy:
  Arm A, C, D:
  100 mg/m²/day by 1-hour IV infusion on days 1,2,3 (total dose 300 mg/m2). On days 1 and 3 start after idarubicin push. For elderly (>65 yrs) patients only two doses of etoposide are foreseen on days 1+3.
  Arm B:
  100 mg/m²/day by 1-hour IV infusion on days 6,7,8 (total dose 300 mg/m2). On days 6 and 8 start after idarubicin push. For elderly (>65 yrs) patients only two doses of etoposide are foreseen on days 6+8.
Drug: Azacitidine — Induction therapy:
  Arm B and C:
  100 mg/m2/day by subcutaneous (SC) injection or 15-minute IV infusion on day 1 to day 5 (total dose 500 mg/m2). Azacitidine is always given prior to idarubicin and etoposide.
  Arm D:
  100 mg/m2/day by SC injection or 15-minute IV infusion on days 4-8 (total dose 500 mg/m2). Azacitidine is always given prior to idarubicin and etoposide.
  Maintenance therapy:
  Arm B, C, D:
  50 mg/m2/day by SC injection on days 1-5 (total dose 250 mg/m2) every 4 weeks. (Maintenance therapy is scheduled for a total duration of 2 years in patients with continuous CR)
  Arms: Arm B; Arm C; Arm D
Drug: Lenograstim — Consolidation therapy:
  subcutaneously daily beginning on day 10 until neutrophil count > 0.5 x 109/l.

SUMMARY:
This is a randomized phase II, four-arm, open-label, multi-center study in adult patients with acute myeloid leukemia (AML) as defined in inclusion/exclusion criteria.

The primary efficacy objective is to evaluate the impact of sequential or concurrent addition of 5-azacytidine to intensive induction chemotherapy with idarubicin and etoposide on the complete remission (CR) rate

Sample size: 336 patients

The treatment duration of an individual patient randomized into one of the three experimental arms (Arm B, C, D) (in case of application of induction, consolidation and maintenance therapy with Azacitidine) is about 30 months.

The treatment duration for patients randomized into the standard arm of the study (Arm A) is about 7 months (in case of application of induction, consolidation and 2-yrs observation as maintenance (without treatment with Azacitidine)).

In case of induction followed by consolidation with allogeneic Stem cell transplantation (SCT) the treatment duration per patient is about 6 months.

Every patient will be followed until month 54 after inclusion into the study. Duration of the study for an individual patient including treatment (induction, consolidation [chemotherapy or allogeneic SCT], maintenance [experimental arm with Azacitidine or observation]) and follow-up period: 54 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected diagnosis of acute myeloid leukemia or related precursor neoplasm, or acute leukemia of ambiguous lineage (classified according to the World Health Organization (WHO) classification)
* Patients considered eligible for intensive chemotherapy
* WHO performance status of ≤ 2
* Age ≥ 18 years. There is no upper age limit.
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis
* Non-pregnant and non-nursing. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration. "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
* Female patients in the reproductive age and male patients must agree to avoid getting pregnant or to father a child while on therapy and for 3 month after the last dose of chemotherapy.
* Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy). Hormonal contraception is an inadequate method of birth control.
* Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy. (while on therapy and for 3 month after the last dose of chemotherapy)
* Signed written informed consent.

Exclusion Criteria:

-AML with other recurrent genetic abnormalities (according to WHO 2008): AML with t(8;21)(q22;q22); RUNX1-RUNX1T1 AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11 AML with t(15;17)(q22;q12); PML-RARA (or variant translocations with other RARA gene fusions)

* AML with NPM1 mutation
* AML with FLT3 mutation
* Performance status WHO >2
* Patients with ejection fraction < 50% by Multi Gated Acquisition Scan (MUGA) or echocardiogram (ECHO scan) within 14 days of day 1
* Organ insufficiency (creatinine >1.5x upper normal serum level; bilirubin, AST or ALP >2.5x upper normal serum level, not attributable to AML; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)
* Uncontrolled infection
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Known positive for Human immunodeficiency virus (HIV)
* Bleeding disorder independent of leukemia
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation.
* No consent for biobanking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2016-10-02 (Actual)

PRIMARY OUTCOMES:
Rates of complete remission (CR) after induction therapy | 56 days
  To evaluate the impact of sequential or concurrent addition of 5-azacytidine to intensive induction chemotherapy with idarubicin and etoposide on the CR rate

SECONDARY OUTCOMES:
Event-free survival | after two years of follow-up
Relapse-free survival | after two years of follow-up
overall survival | after two years of follow-up
days in hospital during each cycle and during the whole intervention | 6 months
Rate of early deaths or hypoplastic deaths (ED/HD) | 56 days
type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 3.0), timing and relatedness of non-hematological toxicity observed during different treatment cycles | 6 months
quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30) | at the end of therapy (in average 6 months) and once a year in the follow-up
  quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, and demographics according to Messerer et al [35].
duration of leukopenia after each consolidation cycle | 42 days
duration of neutropenia after each consolidation cycle | 42 days
duration of thrombocytopenia after each consolidation cycle | 42 days
duration of leukopenia after each induction cycle | 28 days
duration of neutropenia after each induction cycle | 28 days
duration of thrombocytopenia after each induction cycle | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, MD, Principal Investigator — University Hospital of Ulm
Locations (44):
- Austria (5):
  - Universitätsklinikum Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Elisabethinen Krankenhaus Linz, Linz
  - Landeskliniken Salzburg, Salzburg
  - Hanuschkrankenhaus, Vienna
- Germany (39):
  - Universitätsklinikum Charité Berlin, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen Süd, Evangelischs Krankenhaus, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Klinikum Frankfurt-Höchst, Frankfurt
  - Medizinisches Versorgungszentrum Fulda, Fulda
  - Universitätsklinikum Gießen, Giessen
  - Wilhelm-Anton-Hospital Goch, Goch
  - Universitätsklinikum Göttingen, Göttingen
  - Sklepios Klinik Hamburg-Altona, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Hanau, Hanau
  - KRH Klinikum Hannover-Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn, Heilbronn
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Caritas-Krankenhaus Lebach, Lebach
  - Klinikum Lippe, Lemgo
  - Klinikum Lüdenscheid, Lüdenscheid
  - Klinikum der Johannes-Guttenberg-Universität, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Stauferklinikum Schwäbisch-Gmünd, Mutlangen
  - Klinikum rechts der Isar, München
  - Klinikum Passau, Passau
  - Krankenhaus der Barmherzigen Brüder, Regensburg
  - Caritas-Klinik St. Theresia, Saarbrücken
  - Klinikum Stuttgart, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen
  - Helios Klinikum, Wuppertal

REFERENCES:
- [Derived] Schmutz M, Zucknick M, Schlenk RF, Mertens D, Benner A, Weichenhan D, Mucke O, Dohner K, Plass C, Bullinger L, Claus R. Predictive value of DNA methylation patterns in AML patients treated with an azacytidine containing induction regimen. Clin Epigenetics. 2023 Oct 26;15(1):171. doi: 10.1186/s13148-023-01580-z. PMID 37885041